CLINICAL TRIAL: NCT06070038
Title: A Collaborative Theory-based Intervention to Promote Physical Activity Among Sedentary Parents and Their Children
Acronym: ProAct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jyvaskyla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 806/13.00.04.00/2023
Record Dates: First submitted 2023-09-08; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Inactivity/Low Levels of Exercise; Inactivity, Physical
Keywords: Theory of planned behavior; integrated behavior change model; social cognition; physical activity; sedentarism; self-determination theory
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study will consist of a wait list control trial, with one group assigned to receive the intervention immediately, and one group assigned to act as a control group before receiving the intervention after data collection is completed. The model also includes a stopping rule, such that 12-month follow-up data will not be collected if there is no significant effect of the intervention on the primary outcome (i.e. leisure time PA) at the 3-month follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Immediate intervention group. Participants assigned to the immediate intervention group will be delivered materials over a three-month period as a series of four zoom hosted workshops, online content, and a social support group.
  Interventions: Behavioral: Integrated Behaviour Change Based Intervention Materials
- Waitlist Control Group (Other): Wait-List Control Group. Participants in the follow-up group will be delivered intervention materials following the third data collection timepoint.
  Interventions: Behavioral: Integrated Behaviour Change Based Intervention Materials

INTERVENTIONS:
Behavioral: Integrated Behaviour Change Based Intervention Materials — The intervention will be delivered over a three-month period as a series of four zoom hosted workshops, online content, and a moderated social support group. Zoom workshops will last 45 minutes and will target key constructs from the integrated behavior change model. Main topics of the workshops are autonomy Supportive parenting (Week 1), goal setting and outcome beliefs (Week 3), physical activity norms (Week 5), and encouraging self-efficacy and maintenance (Week 8). Following each workshop, participants will receive links to online content that builds on workshop themes, such as messages, worksheets, and reflection tasks. Throughout the trial, participants will be able to participate in social support chat groups to discuss their progress with other members of the intervention group and intervention facilitators.

SUMMARY:
Insufficient physical activity in children and adults is linked to increased risk of physical and mental health conditions. Parents have an important influence on their children's activity, and preliminary aimed at promoting physical activity suggest the family unit as a potentially efficacious means of delivery. However, there is relatively little research examining the efficacy of family interventions aimed at promoting both parents' and children's physical activity. In addition, many family-based interventions are not guided by behavioral theory known to enhance intervention efficacy and reduce variability, and do not target low-active families. This project will therefore develop and test the efficacy of a theory-based behavioral intervention to increase physical activity engagement in low-active children and their parents. The intervention will adopt a randomized waitlist-controlled design with parents and their children allocated to an intervention group that receives theory-based content targeting changes in key behavioral determinants or to a waitlist control group that receives measurement only. The intervention will be delivered to parent-child dyads in a series of four online meetings with a trained facilitator, accompanied by web-based supporting materials, and a moderated social support online chat group. The primary dependent variable will be parents' and children's leisure time physical activity, and secondary outcomes will be device measured physical activity (intervention group only) and measures of key theory-based determinants of physical activity, including autonomous motivation, attitudes, subjective norms, self-efficacy, intentions, and perceived autonomy support. These outcomes will be measured at baseline and at 3, 6, and 12 months post-baseline. Parents and children allocated to the intervention group are expected to exhibit higher levels of physical activity and behavioral determinants. Intervention effects on physical activity change are expected to be mediated by the theory-based determinants, consistent with psychological theory. The project will contribute to research by testing the efficacy of a unique intervention based on behavioral theory expected to be effective in promoting physical activity in low-active parents and their children, and providing guidelines and materials that practitioners in health promotion and public health can use in campaigns and national strategies to promote physical activity in this population.

DETAILED DESCRIPTION:
Low levels of physical activity in adult and youth populations are associated with an increased risk of physical and mental health conditions and reduced quality of life. Conversely, regular activity participation is associated with reduced chronic disease risk and better psychological health and well-being. However, studies indicate that most young people and adults do not achieve recommended levels of physical activity. Physical activity participation also tends to decrease throughout childhood, with steep declines observed during adolescence. Consequently, effective means to promote physical activity participation in child and adult populations are needed. While family-based interventions represent a potentially useful environment for delivering behavioural interventions to promote physical activity in both parents and children, few interventions have been applied in this context. Those that have, tend not to have a strong basis in behavioural theory, often focus on short-term change, and are seldom evaluated systematically.

Within this project, we aim to develop an intervention to promote physical activity in low-active parents and their children. Based on previous research, an integrated model based on multiple theories from behavioural science, particularly social psychology, will guide the development of the intervention in the current project. Specifically, the model draws its predictions from two key behavioural theories: self-determination theory (SDT) and the theory of planned behaviour (TPB), two pre-eminent theoretical approaches that have been applied extensively to predict behaviour and guide interventions in health behaviour contexts.

Evidence suggests that a key approach to family-based behavioural interventions aimed at promoting physical activity in young people and their parents should focus on parent-child dyads, as they provide an efficient means to increase physical activity in both parties. Few studies have systematically evaluated the efficacy of behaviour change methods focused specifically on these kinds of dyad in changing physical activity in family-based interventions and further high-quality evidence is needed. Although the proposed integrated model has generally been used as a basis for interventions in individual contexts, it has not hitherto been adopted as a basis for family-based behaviour change interventions focused on dyads, yet is well placed to be adapted to inform such interventions. The model can also be modified to encompass dyad-focused versions of key determinants identified in the model. For example, the model can be modified to include dyad-based self-efficacy perceptions, a family-based revision of the self-efficacy construct in the model, which reflects perceived confidence in performing the target behaviour together with other dyad members and joint appraisal of goal progress.

ELIGIBILITY:
Inclusion Criteria:

* Parent does not undertake at least 150 minutes of moderate-intensity (or 75 minutes of vigorous-intensity) physical activity each week.
* Child does not undertake at least 60 minutes of moderate-intensity or vigorous-intensity physical activity each day.
* Child is aged between 8 and 12 years old

Exclusion Criteria:

* Parent reports that either they or their child is currently meeting physical activity guidelines at screening.
* Parent states that they or their child has some physical condition that prohibits them from safely participating in physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Godin Leisure time physical activity questionnaire | Assessed at pre-intervention, 3 months (i.e., immediately post intervention), 6 months, and 12 months.
  Self-reported leisure time physical activity as assessed by the Godin Leisure time physical activity questionnaire in all participants. Score range from 0 upwards, with higher scores indicating more leisure time physical activity.

SECONDARY OUTCOMES:
Theory of Planned Behavior - Semantic Differential Attitude Scale | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  Online questionnaires will be administered to all participants assessing their attitudes towards engaging in leisure time physical activity. Attitude will be assessed using semantic differential scale items scored between 1 and 5, where higher scores are indicative of a more positive attitude towards engaging in physical activity. Survey items are drawn from Finnish language scales validated and used in the research team's previous work and available at https://osf.io/rfw2g
Theory of Planned Behavior - Subjective Norms Likert Scale | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  Online questionnaires will be administered to all participants assessing their subjective norms around engaging in leisure time physical activity. Subjective norm will be assessed using Likert scale items scored between 1 and 5, where higher scores are indicative of a belief that others would want them to engage in physical activity. Survey items are drawn from Finnish language scales validated and used in the research team's previous work and available at https://osf.io/rfw2g
Theory of Planned Behavior - Percieved Behavioral Control Likert Scale | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  Online questionnaires will be administered to all participants assessing their percieved behavioral control around engaging in leisure time physical activity. Percieved behavioral control will be assessed using Likert scale items scored between 1 and 5, where higher scores are indicative of a belief that the participant is able to engage in physical activity if they so wished. Survey items are drawn from Finnish language scales validated and used in the research team's previous work and available at https://osf.io/rfw2g
Theory of Planned Behavior - Intention Likert Scale | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  Online questionnaires will be administered to all participants assessing their intentions to engage in leisure time physical activity. Intentions will be assessed using Likert scale items scored between 1 and 5, where higher scores are indicative of participants intentions and willingness to engage in leisure time physical activity in future. Survey items are drawn from Finnish language scales validated and used in the research team's previous work and available at https://osf.io/rfw2g
Self-Determination Theory - Autonomous Motivation Likert Scale | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  Online questionnaires will be administered to all participants assessing their level of autonomous motivation to engage in leisure time physical activity. Autonomous motivationwill be assessed using Likert scale items scored between 1 and 5, where higher scores are indicative of participants desire to engage in physical activity as they are personally motivated to do so. Survey items are drawn from Finnish language scales validated and used in the research team's previous work and available at https://osf.io/rfw2g
Self-Determination Theory - Percieved Autonomy Support Likert Scale | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  Online questionnaires will be administered to all participants assessing their level of percieved autonomy support for engaging in leisure time physical activity. Percieved autonomy support will be assessed using Likert scale items scored between 1 and 5, where higher scores are indicative of participants belief that they are provided with an enviroment allowing for choice and self-determination for physical activity. Survey items are drawn from Finnish language scales validated and used in the research team's previous work and available at https://osf.io/rfw2g
Triaxial Accelerometer Recordings | Assessed at baseline, 3 months (immediately post intervention), 6 months, and 12 months.
  For participants assigned to the immediate intervention group, device measured physical activity will be assessed alongside self-reported activity levels using triaxial accelerometer such as the Hooke AM13 or similar. Triaxial accelerometer data will be used to catagorise the amount of time spend engaged in sedentary behaviors, and light, moderate, and vigerous physical activity. Scores for each sedentary behavior, light physical activity, moderate physical activity, and vigerous physical activity time will be recorded as the average number of minutes each day in which each participant spent engaged in that catagory of activity.
Focus Group Intervention Evaluation Data - Qualitiative Interview | Assessed at 3 months, immediately post intervention.
  For participants in the immediate intervention group, the post-intervention (3-months) online questionnaire will include an option for participants to express their interest in attending a 45-minute exit interview on the intervention process. The interviews will be held via Zoom, and audio recorded to accommodate qualitative thematic analysis.
Resource Use Data | Assessed at 3 months, for the time period covering the intervention.
  For participants in the immediate intervention group, their utilisation of intervention recources will be recorded in the form of the number of sessions attended, number of online materials accessed, and the number of messages or reactions sent to the whataspp group.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Hagger, Principal Investigator — University of Jyvaskyla; Keegan Knittle, Principal Investigator — University of Jyvaskyla
Locations (1):
- The Faculty of Sport and Health Sciences, Jyväskylä, Central Finland, Finland

IPD SHARING:
Plan to Share IPD: Yes
All research components including protocols, materials, de-identified data, and analysis protocols and output, will be publicly shared on a permanent open-access repository (OSF.io).
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data will be uploaded following the conclusion of all data collection.
Access Criteria: Data will be openly available.
URL: https://osf.io/q8a9m/

REFERENCES:
- [Derived] Phipps D, Green WT, Aho R, Kettunen E, Biddle S, Hamilton K, Laukkanen A, Aunola K, Chan DK, Hankonen N, Hassandra M, Karkkainen T, Kykyri VL, Polet J, Rhodes R, Ruiz MC, Saakslahti A, Schneider J, Toivonen HM, Lintunen T, Hagger M, Knittle K. A Web-Based Physical Activity Promotion Intervention for Inactive Parent-Child Dyads: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 21;13:e55960. doi: 10.2196/55960. PMID 38512336